CLINICAL TRIAL: NCT04052100
Title: Cost-effectiveness of a Multimodal Prehabilitation Program in High-risk Patients Undergoing to Lung Resection: A Randomized Clinical Trial
Brief Title: Multimodal Prehabilitation in Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Anael Barberan-Garcia, Principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCB/2018/1138
Record Dates: First submitted 2019-04-05; First posted 2019-08-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Prehabilitation; Exercise training; Physical activity; Nutrition; Cognitive behavioural therapy; Smoking cessation
MeSH Terms: conditions — Lung Neoplasms; Motor Activity; Smoking Cessation | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Patients following the standard preoperative policies of opur institution
  Interventions: Other: Usual care
- Prehabilitation (Experimental): Patients following the standard preoperative policies of opur institution and the multimodal prehabilitation program
  Interventions: Other: Multimodal prehabilitation

INTERVENTIONS:
Other: Usual care — The standard preoperative measures will consist of a recommendation for physical activity and advice on tobacco smoking cessation and reduction of alcohol intake. In addition, patients who suffer from iron deficient anemia will receive intravenous iron and those at risk of malnutrition (Malnutrition Universal Screening Tool ≥2 (www.bapen.org.uk/pdfs/must/must_full.pdf)) or that require weight control for obesity (IMC≥30) will perform a nutrition intervention by a nutritionist.
  Arms: Usual care
Other: Multimodal prehabilitation — The experimental group will also carry out a prehabilitation program consisting in:
  A. A motivational interview to reinforce the patient's motivation and generate a commitment in relation to the objectives of the program.
  B. A physical activity promotion program to increase the number of daily steps of patients, measured by a wristband and a mobile App.
  C. A supervised high-intensity exercise training program. D. An individualized nutritional optimization plan with dietary advice and protein supplementation (if necessary). Educational material and motivational messages will be sent through a mobile App.
  F. Psychological support through weekly Mindfulness sessions (1.5 hours duration). Educational material and motivational messages will be sent through a mobile App.
  E. A smoking cessation program consisting psycho-cognitive therapy combined with pharmacological treatment. Educational material and motivational messages will be sent through a mobile App.
  Other Names: Prehabilitation
  Arms: Prehabilitation

SUMMARY:
This trial aims to assess the impact of a multimodal prehabilitation program in high-risk patients undergoing lung resection surgery.

DETAILED DESCRIPTION:
This trial aims to assess the cost-effectiveness of a multimodal prehabilitation program in high-risk patients undergoing lung resection surgery. Secondary objectives are to evaluate the impact of the intervention on: i) Healthcare resuorces use; ii) clinical outcomes; and, iii) patient's and professionals experience with the program.

The program includes X main interventions: i) A motivational interview; ii) A high-intensity exercise training program; iii) A plan for physical activity incentivation; iv) A nutritional optimization program; v) A psicologichal support program; and, vi) A smoking cessation program.

ELIGIBILITY:
Inclusion Criteria:

1. Forced espiratory volume in the first second (FEV1) and/or estimated postoperative lung diffusion capacity for carbon monoxide < 60%; and/or,
2. American Society of Anesthesiologist (ASA) index 3-4; and/or,
3. Peak oxygen uptake among 10-20 mL/kg/min.

Exclusion Criteria:

1. Non-elective surgery;
2. Metastasic disease;
3. Unestable cardiac or respiratory condition; 4) Cognitive or locomotor limitations precluding the adherence to the program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | During initial hospitalization
  Hospital days of stay

SECONDARY OUTCOMES:
Postoperative complications | During initial hospitalization
  Number and severity of postoperative complications
30-day hospital readmissions | To 30 days after surgery
  Hospital readmissions during the first 30 days after surgery
30-day emergency room visits | To 30 days after surgery
  Emergency room visits during the first 30 days after surgery
Physical activity | Baseline and pre-surgery
  Physical activity measured by the Yale Physical Activity Survey (YPAS) (range 0-126 points (the higher, the better))
Aerobic capacity | Baseline and pre-surgery
  Exercise endurance time achieved in a constant work-rate exercise test in cycle-ergometer
Self-perceived physical status | Baseline and pre-surgery
  Physical status measured by the physical domain of the SF-36 questionnaire (range 0-100 points (the higher, the better))
Self-perceived mental status | Baseline and pre-surgery
  Mental status measured by the mental domain of the SF-36 questionnaire (range 0-100 points (the higher, the better))
Psychological status | Baseline and pre-surgery
  Anxiety and depression levels measured by the Hospital Anxiety and Depression (HAD) questionnaire (range 0-42 points (the lower, the better))
Fat free mass index | Baseline and pre-surgery
  Fat free mass index measured by bioimpedance
PCR | Baseline and pre-surgery
  Blood levels of PCR
ultrasensible PCR | Baseline and pre-surgery
  Blood levels of ultrasensible PCR
TNF-α | Baseline and pre-surgery
  Blood levels of TNF-α
IL-6 | Baseline and pre-surgery
  Blood levels of IL-6
IL-8 | Baseline and pre-surgery
  Blood levels of IL-8
IL-10 | Baseline and pre-surgery
  Blood levels of IL-10
8-isoprostane | Baseline and pre-surgery
  Blood levels of 8-isoprostane
fibrinogen | Baseline and pre-surgery
  Blood levels of fibrinogen
leptin | Baseline and pre-surgery
  Blood levels of leptin
adiponectin | Baseline and pre-surgery
  Blood levels of adiponectin
white cells | Baseline and pre-surgery
  Blood levels of white cells

CONTACTS AND LOCATIONS:
Overall Officials: Anael Barberan-Garcia, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barberan-Garcia A, Navarro-Ripoll R, Sanchez-Lorente D, Moises-Lafuente J, Boada M, Messaggi-Sartor M, Gonzalez-Vallespi L, Montane-Muntane M, Alsina-Restoy X, Campero B, Lopez-Baamonde M, Romano-Andrioni B, Guzman R, Lopez A, Arguis MJ, Roca J, Martinez-Palli G. Cost-effectiveness of a technology-supported multimodal prehabilitation program in moderate-to-high risk patients undergoing lung cancer resection: randomized controlled trial protocol. BMC Health Serv Res. 2020 Mar 12;20(1):207. doi: 10.1186/s12913-020-05078-9. PMID 32164687